CLINICAL TRIAL: NCT00440024
Title: A Single-Blind Study to Assess Benefits of a Controlled Daily Skin Care Regimen on Retinoid Intolerant Patients (Derm 570)
Brief Title: The Effect Of A Controlled Daily Skin Care Regimen On Retinoic Acid Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Dana L. Sachs, MD, Professor of Dermatology, Medical School, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 570
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Sun-Damaged Skin; Retinoid Intolerance
Keywords: Sun-Damaged Skin; Retinoid Intolerance; Tazarotene Cream; Dove facial cleanser; Dove moisturizer
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell A (Experimental): Study controlled daily skin care regimen during 'rest period' consisting of Dove Mild Cleanser, Dove Facial Moisturizer with SPF 15 followed by Tazorac
  Interventions: Drug: Tazorac; Drug: Dove Mild Cleanser; Drug: Dove Facial Moisturizer
- Cell B (Placebo Comparator): Subject controlled normal skin care regimen during 'rest period, followed by study controlled daily skin care regime consisting of Dove Mild Cleanser, Dove Facial Moisturizer with SPF 15 followed by Tazorac
  Interventions: Drug: Tazorac; Drug: Dove Mild Cleanser; Drug: Dove Facial Moisturizer

INTERVENTIONS:
Drug: Tazorac — Tazarotene 0.1% cream applied to the face once daily before bed
  Other Names: Tazarotene
Drug: Dove Mild Cleanser — Ultra mild cleanser: Dove Non-foaming cleansing lotion
  Other Names: Dove Non-foaming Cleanser
Drug: Dove Facial Moisturizer — Moisturizing cream - Dove facial moisturizer with SPF 15

SUMMARY:
Sun-damaged skin, caused by chronic exposure to ultraviolet (UV) light, is characterized by features such as wrinkling, uneven skin color, roughness and brown spots. An effective treatment for sun-damage that is commonly prescribed is topical retinoic acid (RA). However, the major drawback of topical RA use has been frequently observed irritation characterized by redness, dry skin and severe itching. In this study, we examine whether a daily skin care regimen comprised of an ultra mild cleanser and an effective moisturizer can help improve tolerance to RA treatment.

DETAILED DESCRIPTION:
Sun-damaged skin, caused by chronic exposure to ultraviolet (UV) light, is characterized by features such as wrinkling, uneven skin color, roughness and brown spots. An effective treatment for sun-damage that is commonly prescribed is topical retinoic acid. However, the major drawback of topical retinoic acid use has been frequently observed irritation characterized by redness, dry skin and severe itching. In this study, we examine whether a daily skin care regimen comprised of an ultra mild cleanser and an effective moisturizer can help improve tolerance to retinoid treatment.

Subjects for whom retinoid treatment is indicated for sun-damage will be recruited into the study. The retinoid intolerance will be established via prior history (detailed questionnaire) and a 2-week retinoid treatment (Tazarotene 0.1% cream) phase followed by clinical evaluation and determination of retinoid intolerance.

Subjects that exhibit retinoid intolerance will continue with the study. Approximately 30 subjects will be put on a controlled daily skin care regimen during the remainder of the study period while the rest of the subjects will continue their normal skin care habits. The controlled skin care regimen will consist of facial cleansing with a Dove ultra mild emollient cleanser and application of Dove facial moisturizer, used as normal. During this period, subjects will be evaluated to determine reduction of retinoid intolerance symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians between the ages of 40 and 90 with moderate to severe sun-damage on the face who are generally healthy may participate.
* You must demonstrate a previous history of retinoid intolerance (established through prior history and the 2-week retinoid treatment phase of this study).
* Women of childbearing potential must agree to use an accepted form of birth control for the entire duration of the study.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* You may not have used any topical or systemic retinoids in the past 6 months.
* Women who are pregnant or nursing may not participate.
* If you have a history of non-melanoma skin cancer on the face in the past 5 years, you may not participate.
* If you have any history of malignant melanoma you may not participate.
* If you have any other skin condition or facial hair that will interfere with the study evaluations, you may not participate.
* If you have a known sensitivity to any of the ingredients in the study cream or Dove products, you may not participate.
* If you are currently on special daily skin care regimens that include cleansing with Dove, Olay, Aveeno or Cetaphil liquid facial cleansers and using facial moisturizers more than twice a day you may not participate.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Retinoid irritation symptoms | Weeks 6, 8, 12, 16, 20 and 24
Improvement of sun-damage (wrinkling, uneven skin color, roughness and brown spots). | At the end of the study (week 24)

SECONDARY OUTCOMES:
Treatment effects, such as erythema, peeling, itching, and burning/stinging will be evaluated at each study visit. | Weeks 6, 8, 12, 16, 20 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Dana Sachs, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States